CLINICAL TRIAL: NCT03053726
Title: Evaluate the Effectiveness and Safety of Variable Frequency Stimulation Compared With Constant Frequency Stimulation for Patients With Idiopathic Parkinson's Disease（RESTEP Study）
Brief Title: Evaluate the Effectiveness and Safety of Variable Frequency Stimulation Compared With Constant Frequency Stimulation for Patients With Idiopathic Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-025
Record Dates: First submitted 2017-01-22; First posted 2017-02-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Parkinson Disease
Keywords: Variable Frequency Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and the outcomes assessor are blinded in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Variable Frequency Stimulation (Experimental): Subjects in this group received variable frequency stimulation of deep brain stimulation
  Interventions: Procedure: Variable Frequency Stimulation
- Constant Frequency Stimulation (Sham Comparator): Subjects in this group received constant frequency stimulation of deep brain
  Interventions: Procedure: Variable Frequency Stimulation

INTERVENTIONS:
Procedure: Variable Frequency Stimulation — vary the frequency of the stimulation parameter

SUMMARY:
In the VFS paradigm the stimulation frequency was set to alternate between high and low frequencies, where the frequency of stimulation or frequency combinations can be changed instantaneously according to damage of the moment rhythms. Variable frequency stimulation is a novel dynamic therapy which breaks through the existing single high-frequency stimulation paradigms. It is the world's first VFS therapy for the brain.

DETAILED DESCRIPTION:
In advanced stages of PD, motor symptoms and dyskinesia are effectively treated by deep brain stimulation (DBS) targeting the subthalamic nucleus (STN) . Traditionally, in this procedure, stimulation is set to a constant frequency electrical stimulation with the physician programming the parameters of stimulation frequency, pulse width and amplitude, and stimulated patients' brain nuclei with single frequency, single pulse width and single amplitude of the electric stimulation. Indeed, high frequency stimulation (HFS) of the STN provides consistent, long-term improvement of the cardinal signs of PD . However, the treatment effects of HFS on the axial symptoms of PD, specifically FOG can be poor often causing further impairment. While this can be alleviated by using relatively low frequency stimulation (LFS) , major concerns in the clinical application of LFS exist in regards to its duration of therapeutic benefit. Previous studies have shown that LFS of the STN improves the axial motor signs in some PD patients, but a loss of therapeutic efficacy is seen in the short term. Thereafter, patients may present increased tremor, rigidity and bradykinesia, which is often intolerable outweighing the initial benefits of LFS therapy for FOG. As such, a suitable treatment strategy for FOG remains to be established.

Based on previous findings on the relationships between stimulation frequency and movement rhythm regulation in the human body, The National Engineering Laboratory for Neuromodulation, Tsinghua University, proposes a method of variable frequency stimulation (VFS) for aiding movement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients With Idiopathic Parkinson's Disease.
2. ≥18 years,both male and female
3. Patients who under deep brain stimulation
4. MMSE score ≥24
5. H-Y≥2.0 under the medicine off/ constant frequency stimulation state
6. The 14 item of UPDRS-II score ≥1
7. The 15 item of UPDRS-II score ≥2
8. Subjects had an ability to walk ≥ 10 meters independently under the medicine off/ constant frequency stimulation state

Exclusion Criteria:

1. Pregnant women or breastfeeding mothers, or woman who cannot take effective measures to prevent pregnancy.
2. Presence of other diseases affecting walking distance, such as joint disease in lower body, spinal disease, neuropathy, serious heart or lung disease.
3. Diseases seriously affecting health and life, such as tumour, serious liver or kidney diseases etc.
4. Patients with epilepsy etc.
5. Presence of mental disorders or dementia.
6. Patients or their families who cannot comprehend the therapy or patients who are unable to give informed consent voluntarily.
7. Patients whom cannot cooperate well with follow-up requirements.
8. Patients excluded based on the researchers judgement for participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-08-18 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Stand-Walk-Sit | at 3 months compare to baseline
  The total time of patients who complete the Stand-Walk-Sit task

SECONDARY OUTCOMES:
United Parkinson's Disease Rate Scale scores | at 3、6 months compare to baseline
The39-item Parkinson's Disease Questionnaire (PDQ-39) scores | at 3、6 months compare to baseline
The Freezing of Gait Questionnaire (FOG-Q) scores | at 3、6 months compare to baseline
Gait and Falls Questionnaire (GFQ) scores | at 3、6 months compare to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Luming Li, Study Chair — Tsinghua University
Locations (9):
- China (9):
  - Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - General Hospital of PLA, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - Nanjing Brain Hospital Affiliated to Nanjing Medical University, Nanjing
  - Changhai Hospital of Shanghai, Shanghai
  - Huashan hospital, Fudan university, Shanghai
  - The General Hospital of Shenyang Military, Shenyang
  - Second People's Hospital of Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jia F, Zhang J, Wang H, Liang Z, Liu W, Wang X, Liu Y, Guo Y, Ling Z, Cai X, Wu X, Wu J, Lv W, Xu X, Zhang W, Li L. Variable- versus constant-frequency deep-brain stimulation in patients with advanced Parkinson's disease: study protocol for a randomized controlled trial. Trials. 2019 Dec 19;20(1):749. doi: 10.1186/s13063-019-3884-4. PMID 31856908